CLINICAL TRIAL: NCT00557895
Title: Evaluation and Long Term Follow-up of Patients With Allergic and Inflammatory Disorders
Brief Title: Evaluation and Long-Term Follow-Up of Patients With Allergic and Inflammatory Disorders
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960129; 96-I-0129
Record Dates: First submitted 2007-11-10; First posted 2007-11-14 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-06-25

CONDITIONS: Allergy; Asthma; Allergic Rhinitis; Mastocytosis; Atopic Dermatitis; Food Allergy
Keywords: Asthma; Hypersensitivity; Peanut Allergy; Eosinophilic Esophagitis; Eosinophilic Gastroenteritis
MeSH Terms: conditions — Hypersensitivity; Asthma; Rhinitis, Allergic; Mastocytosis; Dermatitis, Atopic; Food Hypersensitivity; Peanut Hypersensitivity; Eosinophilic Esophagitis; Eosinophilic enteropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will evaluate and follow patients with various allergic, hypersensitivity and inflammatory disorders. The protocol is not designed to test new treatments; patients will be managed with standard of care therapies. Participants may be referred to other current NIAID protocols as appropriate or to new studies as they are developed, but will not be required to join another study.

Patients with allergic, hypersensitivity or inflammatory disorders between the ages of 3 years and 80 years may be eligible for this study. Conditions of interest include, but are not limited to, asthma, allergic rhinitis, mastocytosis, atopic dermatitis and food allergy.

Participants will have a medical history and physical examination, plus standard tests for diagnosing and treating their specific disorder. Tests may include routine blood and urine studies, X-rays or other imaging studies, allergy skin tests and lung function tests. Blood samples may be collected for research on immune system cells and other substances involved in immune function. Generally, about 2 to 6 tablespoons will be drawn at a time, but no more than 16 ounces will be collected over a 6-week period.

NIH does not provide emergency medical treatment or treatment for other, unrelated conditions the patient may have. Therefore, patients must maintain a personal physician for these purposes.

DETAILED DESCRIPTION:
Allergic, hypersensitivity and inflammatory disorders, including but not limited to asthma, allergic rhinitis, mastocytosis, atopic dermatitis and food allergy are exceedingly common disorders. The pathogenesis of these various disorders are being investigated under a number of Laboratory of Allergic Diseases clinical research protocols. This protocol is an evaluation and long term follow-up protocol of such disorders, for the purposes of maintaining a group of patients on which LAD investigators draw for our other various protocols. The patients admitted under this protocol also provide training and experience for members of the NIAID Allergy and Immunology fellowship training programs.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males and females ages 3 years to 80 years.

Allergic, hypersensitivity or inflammatory diseases.

Willingness to participate in clinical protocols when appropriate.

Subjects must maintain a private physician for non-protocol related medical complaints and for emergency medical treatment required for these or other of their disorders.

EXCLUSION CRITERIA:

Unacceptably poor compliance which, in the opinion of the investigator, would interfere with one's ability to study or provide quality medical care for the patient.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 1996-08-26; Study Completion 2019-06-25

PRIMARY OUTCOMES:
The protocol serves to evaluate and provide long term follow up of patients with allergic, hypersensitivity and inflammatory disorders for the purposes of maintaining a group of patients from which LAD investigators may draw for other protocols ... | The outcome is assessed over the time the protocol is active as described elsewhere.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly D Stone, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Prussin C, Lee J, Foster B. Eosinophilic gastrointestinal disease and peanut allergy are alternatively associated with IL-5+ and IL-5(-) T(H)2 responses. J Allergy Clin Immunol. 2009 Dec;124(6):1326-32.e6. doi: 10.1016/j.jaci.2009.09.048. PMID 20004787